CLINICAL TRIAL: NCT04443998
Title: Evaluation of Bone Reduction Forceps in Reducing Mandibular Fracture
Brief Title: Mandibular Fracture Reduction Using Bone Reduction Forceps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mandibular fracture reduction
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone reduction forceps (Experimental)
  Interventions: Device: Bone reducion forceps

INTERVENTIONS:
Device: Bone reducion forceps — Repositioning forceps provide a more accurate anatomical reduction and higher pre-compression can be achieved compared to IMF or manual reduction

SUMMARY:
Different methods have been used in reducing mandibular fractures. Bone reduction forceps provides precise reduction and stabilize mandibular fracture segments.

DETAILED DESCRIPTION:
The aim of this study is to evaluate clinically and radiographically the effect of using bone reduction forceps in the reduction of isolated mandibular fractures.

10 patients complaining of isolated mandibular fractures in need of open reduction and internal fixation underwent reduction using bone reduction forceps.

The patients followed up clinically after 1 and 2 weeks, 1, 3, and 6 months postoperatively. Radiographic evaluation will be performed by computed tomography (CT) preoperatively, and cone-beam computed tomography (CBCT) will be done after 3 and 6 months

ELIGIBILITY:
Inclusion criteria

* Adult patients aged from 20 to 45 years will be included.
* Patients suffered from recent and uninfected.
* Patients with isolated mandibular fractures.

Exclusion criteria

* Medically compromised patients that will be not fit for surgery.
* Edentulous patients.
* Non-displaced
* Comminuted fracture with bone loss
* Old fracture, more than 3 weeks

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-08-18 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in radiodensitometric measurements | at 3rd, 6th months
  cone-beam computerized tomograms (CBCT) used to analyze the mean bone density at the site of fracture
change in maximal mouth opening | 1 week, 2 weeks, 1 month, 6 weeks, and 3 months
  maximal interincisal opening between maxillary and mandibular central incisors.
change in occlusion | 1 week, 2 weeks, 1 month, 6 weeks, and 3 months
  Any occlusal disturbance including open bite or improper tooth contact will be recorded
change in pain level | 1 week, 2 weeks, 1 month, 6 weeks, and 3 months
  Pain: will be measured on Visual Analogue Scale (VAS). The patients will be asked to rate their postoperative pain on a 4-point scale (0= none, 1= slight, 2= moderate, 3- severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt